CLINICAL TRIAL: NCT05045898
Title: Effects of Textured Insoles Used in Addition to Foot Massage Application on Balance, Sensation, Foot Functions, Physical Activity and Quality of Life in Individuals Diagnosed With Rheumatoid Arthritis
Brief Title: Textured Insoles and Foot Massage in Individuals Diagnosed With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gamze Pala, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021 - 848
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: plantar massage; textured insoles; balance; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): plantar massage
  Interventions: Other: plantar massage
- Intervention group (Experimental): plantar massage and textured insoles
  Interventions: Other: plantar massage; Other: textured insoles

INTERVENTIONS:
Other: plantar massage — The patients will be given a classical massage, known as Swedish massage, consisting of euflorage and petrissage. While the patient is lying in the supine position, a classical massage will be applied to the plantar face, dorsum and toes of both feet, which will take approximately 20 minutes in total. It will last for 6 weeks, 3 days a week.
Other: textured insoles — Textured insoles will be prepared in accordance with the principles stated by Waddington et al. in 2003. In the studies of Waddington et al., ethyl vinyl acetate (EVA) textured insoles with 4 hemispherical protrusions per cm² were used. The height of each hemispherical protrusion from the EVA floor is 2 mm; The height of the insoles from the ground is 3 mm.
  The textured insoles will be prepared by an orthotic prosthesis center by cutting the EVA layer with the above-mentioned features in accordance with the patient's shoe/home shoe insoles and placing them on the shoe/home shoe insoles. Insoles will be provided free of charge to patients. Patients will be asked to wear their shoes/house shoes with insoles while performing activities inside and outside the home for 6 weeks.
  Arms: Intervention group

SUMMARY:
The aim of this study is to determine and compare the effects of using textured insoles and plantar massage on balance in patients with rheumatoid arthritis. Patients diagnosed with rheumatoid arthritis will be divided into two groups. In the first group the patients will be given plantar massage; in the second group, both plantar massage will be applied and the patients will use textured insoles in their indoor and outdoor activities. Plantar massage will be applied by the physiotherapist 3 days a week for 6 weeks; textured insoles will also be used for 6 weeks. All patients will be asked to complete the questionnaires, which assessed foot functionality, physical activity levels and quality of life. After each patients completed the questionnaire, the physiotherapist will perform plantar sensory and balance assessment. All assessments will be made before, after and 8 weeks after treatment.

DETAILED DESCRIPTION:
In the solution of balance problems in rheumatoid arthritis (RA), successful results can be obtained with the correct sensory inputs from the sole of the foot. Even after 5 minutes of application with plantar massage, which is one of these methods, it has been observed that there is an improvement in balance reactions. Textured insoles are also one of the methods used to improve balance with the right sensory input. Both methods increase cutaneous receptor activity and ankle proprioception by providing increased afferent information; As a result of these effects, postural sway decreases, balance can be achieved on a narrower support surface, and postural control increases. Although the positive effects of plantar massage and textured insoles on balance are known, there are no studies in which these methods are used in RA patients. In our study, we aimed to determine and compare the effects of plantar massage, which provides short-term afferent input, and the use of textured insoles, which provide long-term afferent input, on balance in RA patients. For these purposes, plantar massage will be applied to one group, and plantar massage will be applied to the other group and textured insoles will be used. In this way, the effects on the balance will be observed and compared.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Being diagnosed according to the American College of Rheumatology (ACR)/EULAR 2010 rheumatoid arthritis diagnostic criteria

Exclusion Criteria:

* Having an orthopedic or neurological disease that may cause balance and sensory impairment
* Using drugs that may cause balance and sensory disorders
* Having undergone lower extremity surgery
* Having a neurological problem that may cause hearing or vision impairment
* Having a communication problem
* Having a history of major psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Foot Function Index | Before treatment.The activity limitation subscale includes 5 items and evaluates activity limitations due to foot problems. Each item is scored between 0 and 10. A high score indicates a high degree of disability.
  The feet are flexible structures of bones, joints, muscles, and soft tissues that let us stand upright and perform activities like walking, running, and jumping. Foot functions will be evaluated with the Foot Function Index.
International Physical Activity Questionnaire Short Form | Before treatment. After scoring, physical activity levels are classified as physically inactive (inactive), low physical activity level (minimally active), and adequate physical activity level (very active).
  Physical activity refers to all movement including during leisure time, for transport to get to and from places, or as part of a person's work. The physical activity levels of the patients will be evaluated with the International Physical Activity Questionnaire Short Form.
Health Assessment Questionnaire | Before treatment. The health assessment questionnaire consists of 20 questions, each question is scored between 0-3. A high score indicates poor functional status.
  Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time. health-related quality of life will be assessed by Health Assessment Questionnaire.
Plantar sensory assessment | Before treatment. The score of the thinnest monofilament felt will be recorded.
  Light touch-pressure and functional sense assessment. plantar sense will be performed by a physiotherapist with Semmes-Weinstein monofilament test and two-point discriminator.
Balance | Before treatment. With the tests, the ability of the patients to maintain the center of balance, to move the center of gravity between the support surfaces of the body and to control it will be evaluated.
  A state of equilibrium or parity characterized by cancellation of all forces by equal opposing forces. Balance assessment will be done by the physiotherapist with the Biodex Balance System.
Foot Function Index | After 6 weeks. The activity limitation subscale includes 5 items and evaluates activity limitations due to foot problems. Each item is scored between 0 and 10. A high score indicates a high degree of disability.
  The feet are flexible structures of bones, joints, muscles, and soft tissues that let us stand upright and perform activities like walking, running, and jumping. Foot functions will be evaluated with the Foot Function Index.
International Physical Activity Questionnaire Short Form | After 6 weeks. After scoring, physical activity levels are classified as physically inactive (inactive), low physical activity level (minimally active), and adequate physical activity level (very active).
  Physical activity refers to all movement including during leisure time, for transport to get to and from places, or as part of a person's work. The physical activity levels of the patients will be evaluated with the International Physical Activity Questionnaire Short Form.
Health Assessment Questionnaire | After 6 weeks. The health assessment questionnaire consists of 20 questions, each question is scored between 0-3. A high score indicates poor functional status.
  Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time. health-related quality of life will be assessed by Health Assessment Questionnaire.
Plantar sensory assessment | After 6 weeks. The score of the thinnest monofilament felt will be recorded.
  Light touch-pressure and functional sense assessment. plantar sense will be performed by a physiotherapist with Semmes-Weinstein monofilament test and two-point discriminator.
Balance | After 6 weeks. With the tests, the ability of the patients to maintain the center of balance, to move the center of gravity between the support surfaces of the body and to control it will be evaluated.
  A state of equilibrium or parity characterized by cancellation of all forces by equal opposing forces. balance assessment will be done by the physiotherapist with the Biodex Balance System.
Foot Function Index | After 14 weeks. The activity limitation subscale includes 5 items and evaluates activity limitations due to foot problems. Each item is scored between 0 and 10. A high score indicates a high degree of disability.
  The feet are flexible structures of bones, joints, muscles, and soft tissues that let us stand upright and perform activities like walking, running, and jumping. Foot functions will be evaluated with the Foot Function Index.
International Physical Activity Questionnaire Short Form | After 14 weeks. After scoring, physical activity levels are classified as physically inactive (inactive), low physical activity level (minimally active), and adequate physical activity level (very active).
  Physical activity refers to all movement including during leisure time, for transport to get to and from places, or as part of a person's work. The physical activity levels of the patients will be evaluated with the International Physical Activity Questionnaire Short Form.
Health Assessment Questionnaire | After 14 weeks. The health assessment questionnaire consists of 20 questions, each question is scored between 0-3. A high score indicates poor functional status.
  Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time. health-related quality of life will be assessed by Health Assessment Questionnaire.
Plantar sensory assessment | After 14 weeks.The score of the thinnest monofilament felt will be recorded.
  Light touch-pressure and functional sense assessment. plantar sense will be performed by a physiotherapist with Semmes-Weinstein monofilament test and two-point discriminator.
Balance | After 14 weeks. With the tests, the ability of the patients to maintain the center of balance, to move the center of gravity between the support surfaces of the body and to control it will be evaluated.
  A state of equilibrium or parity characterized by cancellation of all forces by equal opposing forces. balance assessment will be done by the physiotherapist with the Biodex Balance System.

CONTACTS AND LOCATIONS:
Overall Officials: Deran Oskay, Prof, Principal Investigator — Gazi University; Abdurrahman Tufan, Prof, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qiu F, Cole MH, Davids KW, Hennig EM, Silburn PA, Netscher H, Kerr GK. Effects of textured insoles on balance in people with Parkinson's disease. PLoS One. 2013 Dec 12;8(12):e83309. doi: 10.1371/journal.pone.0083309. eCollection 2013. PMID 24349486
- [Background] Wikstrom EA, Song K, Lea A, Brown N. Comparative Effectiveness of Plantar-Massage Techniques on Postural Control in Those With Chronic Ankle Instability. J Athl Train. 2017 May 23. doi: 10.4085/1062-6050.52.4.02. Online ahead of print. PMID 28535097
- [Background] Waddington G, Adams R. Football boot insoles and sensitivity to extent of ankle inversion movement. Br J Sports Med. 2003 Apr;37(2):170-4; discussion 175. doi: 10.1136/bjsm.37.2.170. PMID 12663362